CLINICAL TRIAL: NCT07063849
Title: A Pilot Study of the Effects of Pre-Existing Immunity on Influenza A/Texas/71/2017 (H3N2) Virus Shedding After Human Challenge in Healthy Participants
Brief Title: Pilot Influenza Challenge Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Hoft, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Daniel Hoft, MD, PhD, Professor of Internal Medicine, St. Louis University
Organization: St. Louis University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SLU-25-001
Record Dates: First submitted 2025-06-16; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-05

CONDITIONS: Influenza
Keywords: CHIM; Challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): One dose of RG-A/Texas/71/2017 Influenza Virus
  Interventions: Biological: A/Texas

INTERVENTIONS:
Biological: A/Texas — Live Influenza Virus RG-A/Texas/71/2017 H3N2 Dose: 1.0 mL (0.5mL per nostril) of approximately 1x10^6 TCID50 Administered intranasally by atomizer device Challenge virus will be administered once on Day 1

SUMMARY:
This is a research study to understand what happens when a person is infected with influenza ("flu") and how the body controls the infection. Healthy participants (challenge) will be infected with a strain of flu (H3N2), and followed to see what symptoms occur and when they occur. Blood will be drawn and nasopharyngeal (NP) swabs will be collected before participants are infected to understand if having antibodies can protect participants from flu infection or lead to a milder flu illness. Blood will also be drawn and NP swabs collected after participants are infected to understand how and when the body's immune response to flu occurs. Participants will also breathe through a device for virus collection every other day.

Participants will be screened during one or more visits and will stay in the inpatient challenge unit for at least 10 days, maybe longer. Participants will complete a FLU PRO Diary Card daily. Blood will be drawn before the challenge and on Days 2, 4, and 8 while in the inpatient unit. NP samples will be taken every day to check for viruses and on certain days, immune responses such as antibodies. If on Day 8 (7 days after the challenge) the participant still has flu virus, medicine will be offered to treat the flu and the participant will be asked to stay in the challenge unit until NP swabs are negative for 2 consecutive days. Once the participant is discharged from the challenge unit, they will be asked to return to the clinic for 3 more visits. At the end of the study will be a final phone call.

DETAILED DESCRIPTION:
This experimental pilot study is designed to develop methods to analyze viral complexity shed after experimental human infection with influenza A virus, a necessary first step in the development of mucosal transmission models. While the initial influenza CHIM study at SLU employed an H1N1 influenza strain, in this study, an H3N2 strain will be used. Data reported from the first-in-human, dose-finding study for the DMID- and CIVICs-developed, RG-A/Texas/71/2017 (H3N2). Similarly, while the use of different clinical scoring rubrics prevents direct comparisons, illness observed during DMID 18-0010 was reported to be very mild, and lacked a sham inoculum comparator group, but the raw data are not available for review. In contrast, with RG-A/Texas/71/2017 (H3N2), participants reported a mean cumulative MJS of 25.8 (range 18.3 to 34.1) from day 2 through day 8; the MJS ranges from 0 to 36 for each measurement. In contrast, both of the sham inoculated participants had a cumulative MJS of 1.0. These observations are consistent with comparisons between H1N1 and H3N2 during naturally acquired infection. Thus, the H3N2 CHIM may be more amenable to studies of shed virus and mucosal immunity, and to provide a wider dynamic range of influenza illness against which to test vaccine and treatment countermeasures in the future. This study will examine the genetic diversity of shed influenza virus particles in small (<5µm) versus large (≥5µm) exhaled particles, as well as in nasopharyngeal swab samples, and compare the viral diversity in these specimens stratified by baseline serum microneutralization titer and nasopharyngeal mucosal IgA titers. While this is a small, exploratory study, not powered for statistical significance of endpoints, the aim is to develop the methods necessary for future, larger scale studies to apply this practical knowledge to further understand mucosal immune correlates of protection against influenza A disease. This understanding will be valuable for the development and testing of new influenza vaccines that better leverage mucosal immunity against influenza infection and transmission.

This is a CHI study of Influenza RG- A/Texas/71/2017 (H3N2) influenza, clade 3C3a virus to assess clinical response, immunological response, and safety. The study population will be healthy participants (male and non-pregnant, non-breastfeeding females) between the ages of 18 to 45, inclusive. Up to 12 participants will receive H3N2 virus CHI. Clinical manifestations, viral shedding, and immunological responses will be characterized.

Influenza RG-A/Texas/71/2017 (H3N2) influenza, clade 3C3a virus CHI will be performed using a 12 mL dose of approximately 1.86 x10^6 TCID50/mL, which has been shown to induce 60% or higher rates of MMID. The primary objective of the study will be to evaluate the association of MMID post-challenge and pre-existing virus-specific HAI titers in healthy participants. MMID is defined as the presence of both of the following, assessed through Day 8:

* Viral shedding detected by any approved positive RT-PCR assay from a NP swab, and
* Any one or more of the following symptoms or signs or laboratory findings, as related to the study agent; Arthralgia, Chest tightness, Chills, Conjunctivitis, Nasal congestion, Sinus Congestion, Coryza, Decreased appetite, Diarrhea, Dry Cough, Dyspnea/Shortness of Breath, Fatigue/Tiredness, Fever (>38.0°C), Headache, Lymphopenia (<1000 cells/mL), Myalgia, Nausea, Oxygen Saturation Decrease by ≥3% from baseline, Productive Cough, Rhinorrhea, Sore Throat, and Sweats.

During Study Days -30 to -3 (Screening Period), participants will provide informed consent to participate in this study. They will undergo a review of medical history, physical examination by a study physician, and screening laboratory tests. During this period, participants will also have a posteroranterior (PA) and Lateral chest X-ray (CXR), and a baseline 12-lead ECG.

After screening, eligible participants will be admitted to an inpatient challenge unit (Day -2). Up to twelve participants will be enrolled of which up to 6 participants will have H3N2 challenge titers <40 and up to 6 participants will have H3N2 challenge titers >40. The plan is to enroll participants with the broadest range of MN titers. Based on the results of the MN titers, participants may be healthy but may not be enrolled. Backup participants may be admitted into the inpatient unit to ensure sufficient number of volunteers undergo CHI, given the potential for drop-outs, presence of new exclusionary criteria, and/or pre-challenge evidence of viral respiratory infection among participants. A review of eligibility criteria, and baseline clinical assessments, safety blood tests, influenza virology, and immunology tests will be performed and the participants will have approximately a 48-hour window to decide if they would like to drop out of the study and leave the inpatient unit before CHI. Participants must have no evidence of a respiratory viral infection as determined by multiplex respiratory virus RT-PCR assay testing prior to CHI (positive results prior to CHI will exclude the subject from the challenge, and additional participants may serve as replacements). On Day -1, participants will be trained on the influenza patient related outcomes Flu-PRO Survey Instrument and Validation Diary.

On Day 1, eligibility and clinical status will be reviewed. If criteria for proceeding with challenge are met, participants will receive A/Texas/71/2017 (H3N2), clade 3C3a CHI. 0.5 mL of RG-A/Texas/71/2017 (H3N2) influenza, clade 3C3a will be delivered in each nostril of a recumbent participants per study SOP. Backups will be discharged from the inpatient unit prior to challenging other participants if not needed to replace ineligible participants or participants declining to proceed with CHI.

After CHI, participants will complete daily self-assessments using the Flu-PRO Survey Instrument and Validation Diary through 14 days post-challenge to generate a symptom severity score. Participant clinical status will be monitored closely. Safety labs will be performed at scheduled times. Participants will undergo scheduled blood draws, and nasal swab collections for immunology and virologic laboratory testing. Quantitative and qualitative evaluation of influenza will be done after CHI on Day 7. Participants will also undergo qualitative evaluations for evidence of influenza by multiplex respiratory virus RT-PCR assay. Participants will speak/breathe into the PathoSift Pro which is a Bioaerosol Sampler device for 15-30 minutes every other day while in the confinement unit to collect airborne viruses. Participants will remain blinded to the results of their respiratory virus testing until they meet discharge criteria. An ECG will be performed at Day 6 on all participants, and as clinically indicated at any other time.

Following CHI, participants will remain in the inpatient unit for a minimum of seven additional days and will be discharged only if 1) they have two consecutive negative influenza tests (that are performed on days 7 and 8) for influenza A using a multiplex respiratory virus assay (BIOFIRE® FILMARRAY® or Luminex xTAG®), AND 2) have been afebrile (<38.0°C), have a room air Saturation of Peripheral Oxygen (SpO2) ≥95 and have been clinically and hemodynamically stable for at least 48 hours. In addition, participants may have residual and/or resolving symptoms of influenza illness. It is expected that most participants will shed the challenge virus for three to five days post exposure.

If participants are still shedding virus on Day 8, they will remain in the challenge unit, be offered one dose of baloxavir marboxil (a full treatment course), and they will continue to have NP swabs tested daily until there are two negative influenza tests performed on consecutive days and meet clinical discharge criteria described above.

Any participant who develops serious related or unrelated signs or symptoms during inpatient stay will receive appropriate and as clinically necessary escalation of care (e.g., cardiologist consultation for cardiac symptoms or transfer for evaluation at the Emergency Department). Any participant who experiences complications or sequelae due to CHI will be followed until resolution and/or stable, and will be referred for appropriate specialized care as clinically necessary. All participants will be followed for approximately 90 days post-challenge. Additional follow-up will be performed at in-person Visits 9 (Day 15), 10 (Day 29) and 11 (Day 61). Participants will also undergo scheduled blood draws and nasopharyngeal (NP) swabs for immunology and virologic laboratory testing during this follow up period. A final follow-up by telephone will occur on Visit 12 (Day 91).

ELIGIBILITY:
Inclusion Criteria

Participants eligible to participate in this study must meet all of the following inclusion criteria:

1. Provide written informed consent prior to initiation of any study procedure.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Agree to remain an inpatient for at least seven days after challenge, AND until they have no virus shedding,1 determined by qualitative RT-PCR for a minimum of two consecutive days post-challenge 1For a minimum of seven days post-challenge (Study Day 8).
4. Healthy2 males and non-pregnant, non-breastfeeding females3 aged ≥18 and ≤45 years of age, inclusive, at enrollment.

2Good health is defined in inclusion criteria #10. 3Females participants of childbearing potential must agree to have a serum pregnancy test at screening, a urine pregnancy test before CXR performed (if more than 7 days have passed between CXR and serum pregnancy test), and a urine pregnancy test upon admission to the inpatient unit prior to CHI, and results must be negative.

5. Women of childbearing potential4 must agree to use or have practiced true abstinence5 or use at least 1 acceptable primary form of contraception6,7 These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to participants in a same sex relationship).

4Not of child- bearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement with history of documented radiological confirmation test at least 90 days after the procedure).

5True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

6Acceptable forms of primary contraception include intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products monogamous relationship with a vasectomized partner who has been vasectomized for180 days or more prior to the subject receiving the influenza challenge virus.

7Must use at least one acceptable primary form of contraception for at least 30 days prior to admission and at least one acceptable primary form of contraception during the remainder of the study.

6. Non-habitual smoker8 of tobacco, or marijuana. 8Non-habitual smokers are those who smoke no more than four cigarettes, other tobacco products, vaping (e-cigarettes) or marijuana in a week for more than three months and agree not to smoke cigarettes, other tobacco products, e-cigarettes and/or marijuana products during participation in the study.

7. No self-reported or known history of alcoholism or drug use within the last 30 days and agrees to abstain from alcohol and drugs9 for at least one week before admission and throughout the inpatient period.

9 including forms of marijuana not included in criterion 6 8. Negative drug urine toxicology result on screening (i.e., amphetamines, cocaine, and opiates). and on admission to the challenge unit (i.e., amphetamines, cocaine, and opiates).

9. Agree not to use the listed10 prescription or over-the-counter medications within 7 days prior to inpatient stay and through inpatient stay, unless approved by the investigator.

10Oseltamivir, zanamivir, peramivir, baloxavir marboxil, amantadine (generic) and rimantadine (Flumadine and generic), aspirin, intranasal steroids, decongestants, antihistamines, and other non-steroidal anti-inflammatory drugs (NSAIDs).

10. In good health11 and not have clinically significant medical, psychiatric, chronic or intermittent health conditions including those listed in Exclusion Criteria.

11Good health, as determined by medical history, medication use and physical examination to evaluate ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would not affect the assessment of the safety of participants or the immunogenicity of challenge. These medical diagnoses or conditions should be stable for the last 90 days (no hospitalizations, emergency room (ER) or urgent care for condition (excluding musculoskeletal conditions) and not listed in Exclusion Criteria (Section 5.1.2). Participants may be on medications only if the condition or disease is stable and not deteriorating, if the medical intervention (such as device or medication) was not available during the maximal inpatient period of time, medications are not listed in the Exclusion Criteria (Section 5.1.2.) and pose no additional risk to subject safety or assessment of adverse events. This also includes no change in prescription medication, dose or frequency as a result of new symptoms or deterioration of the medical diagnosis or condition in the 90 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome (e.g., lowering of the dosage or frequency), as determined by the site principal investigator (PI) or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572, will not be considered a deviation of this inclusion criterion.

11. Does not have an ongoing symptomatic condition12 for which subject has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan.

12e.g., ongoing fatigue without a diagnosis for symptom. 12. Vital signs as follows13: 13pulse is 47 to 99 beats per minute, inclusive; systolic blood pressure is 85 to 139 mmHg, inclusive; diastolic blood pressure is 55 to 89 mmHg, inclusive; SpO2 >95%; RR<18; oral temperature is less than 100.0°F.

13. Eligibility laboratory values (WBC, Absolute Lymphocyte Count, Hgb, PLTs, ALT and Cr) are within acceptable parameters.

14. Body mass index (BMI) >18.5 and <35 kg/m2 at screening. 15. Other screening tests (ECG and CXR) are within normal reference range or not deemed clinically significant by the PI or appropriate sub-investigator14 14Designated clinician licensed to make medical diagnoses and listed on the Form FDA 1572 16. H3N2 Challenge virus MN titer done in SLU VTEU research lab during screening to allow selection for enrollment of subjects with the broadest range of pre-existing H3N2 immunity.

17. Negative test for HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV) at screening blood draw.

18. Negative respiratory virus panel by BIOFIRE® FILMARRAY® respiratory panel by bioMérieux or by Luminex xTAG® on Day -2, and Day -1.

Exclusion Criteria

Participants eligible to participate in this study must not meet any of the following exclusion criteria:

1. Female subject who has a positive pregnancy test on screening or admission, is breastfeeding or planning to become pregnant from 30 days prior to challenge through the end of the study.
2. Presence of self-reported or medically documented significant medical or psychiatric condition(s)15 15Significant medical or psychiatric conditions include but are not limited to:

   1. Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications15 currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years 16Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.
   2. Presence of any febrile illness or symptoms suggestive of a respiratory infection within two weeks prior to CHI.
   3. Cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
   4. Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barre syndrome, encephalomyelitis or transverse myelitis).
   5. Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell carcinoma of the skin, which is allowed.
   6. An autoimmune disease.
   7. An immunodeficiency of any cause.
   8. A history of diabetes.
3. Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness17- 17Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 12-month period prior to screening. Low dose topical and intranasal steroid preparations used for a discrete period of time are permitted (Section 7.1).
4. Known allergy or intolerance to treatments for influenza (including but not limited to oseltamivir, baloxavir marboxil, acetaminophen).
5. Known allergy to two or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
6. Known allergy to excipients in the challenge virus inoculum.
7. Receipt or planned receipt of any investigational drug/investigational vaccine/licensed vaccine within 30 days prior to the date of CHI.
8. Prior enrollment in any influenza virus challenge study.
9. Currently enrolled in any investigational study or intends to enroll in such a study within the ensuing study period.
10. Receipt of any influenza vaccine six months prior to challenge or plans to receive influenza vaccine within 60 days post-challenge.
11. History of a previous severe allergic reaction of any kind with generalized urticaria, angioedema, or anaphylaxis.
12. Receipt of blood or blood products during the six months prior to the planned date of challenge.
13. History of blood donation during the two months prior to the planned date of challenge and or plans to donate blood for the duration of the study.
14. Any condition, to include medical and psychiatric conditions, that in the opinion of the Investigator, might interfere with the safety of the subject and/or study objectives.
15. Known close contact with anyone known to have influenza 7 days prior to challenge.
16. Acute medical condition with new prescription medication use in the last 30 days.
17. Significant abnormality altering the anatomy of the nose/nasopharynx18 clinically significant nasal deviation, or nasal/sinus surgery within 180 days prior to challenge.

18including significant nasal polyps. 18. History in the last five years of chronic or frequent intermittent sinusitis.

19. Recent history (180 days) of epistaxis or anatomic or neurologic abnormality impairing the gag reflex or contributing to aspiration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) and Serious Adverse Events (SAE) during inpatient challenge | Post-challenge Day 1 through Day 8
Frequency of AE and SAE post-inpatient discharge | Thoughout the duration of the study (approximately three months post challenge)
FLU-PRO symptomatic scoring of clinical symptoms twice daily | Day 2 through at least Day 8 after challenge
H3N2-specific polymerase chain reaction (PCR) on nasopharyngeal (NP) samples daily | Day 2 through at least Day 8 post-challenge
H3N2 viral loads as assessed by quantitative reverse transcription polymerase chain reaction (qRT-PCR). | Days 2, 4, 6, and 8 post challenge
H3N2 viral clonotypic complexity by Next-Gen sequencing of NP and exhaled breath samples. | Days 2, 4, 6, and 8 post challenge
Studies of biologically relevant mutations in the H3N2 viral genome post-challenge discovered by Next-Gen sequencing of NP and exhaled breath samples | Days 2, 4, 6, and 8 post challenge
Relative abundance of live H3N2 virus shed in exhaled breath within droplets (diameter greater than or equal to 5 microns) and aerosols (diameter less than 5 microns) | Days 2, 4, 6, and 8 post challenge
H3N2 viral loads as assessed by median tissue culture infective dose (TCID50) assays | Days 2, 4, 6, and 8 post challenge

SECONDARY OUTCOMES:
Proportions positive for virus shed into NP swabs on different days post-challenge using qRT-PCR. | From baseline (Day -2 or -1) and daily from Day 2 through Day 8
Baseline and post-challenge hemagglutination inhibition (HAI) and microneutralization (MN) antibody Geometric Mean Titers (GMTs) from serum | Baseline (Day -2), and Days 8, 29, and 61.
Percentage of participants achieving HAI and MN seroconversion (either a pre-challenge titer <1:10 and a post-challenge titer of greater than or equal to 1:40 or a pre-challenge titer of greater than or equal to 1:10 and a four-fold rise post-challenge | Baseline (Day -2), and on Days 8, 29, and 61
Baseline and post challenge H3HA-specific secretory GMTs by ELISA in NP swab samples | Baseline (Day -2), and on Days 8, 29, and 61
Spearman correlations between HAI/MN titers pre-challenge and FLU PRO scoring levels post-challenge | Day 1 prior to the challenge through Day 14
Spearman correlations between HAI/MN titers pre-challenge and Area Under the Curve (AUC) of total viral shedding over time post-challenge by qRT-PCR | Baseline (Day -2), and on Days 8, 29, and 61
Spearman correlations between baseline HAI/MN titers and level of clonotypic complexity shed on exhaled breath | Baseline (Day -2) and on Days 2, 4, 6, and 8 post challenge
Spearman correlations between baseline HAI/MN titers and numbers of mutations accumulating in viral strains shed in exhaled breath post challenge | Baseline (Day -2) and on Days 2, 4, 6, and 8 post challenge
Spearman correlations between H3HA-specific secretory IgA (sIgA) GMTs pre-challenge and FLU-PRO scoring levels post-challenge | Baseline (Day -2), and through Day 14 post-challenge
Spearman correlations between baseline H3HA-specific sIgA titers and AUC of total viral shedding over time post-challenge by qRT-PCR. | Baseline (Day -2) pre-challenge, and through Day 61 post-challenge
Spearman correlations between baseline H3HA-specific sIgA titers and level of viral clonotypic complexity shed in exhaled breath post-challenge | Day -2 pre-challenge and Days 2, 4, 6, and 8 post-challenge
Spearman correlations between baseline H3HA-specific sIgA titers and numbers of mutations accumulating in viral strains shed in exhaled breath post-challenge | Baseline (Day -2) pre-challenge and Days 2, 4, 6, and 8 post-challenge
Peak magnitude of virus shed into NP swabs post-challenge using qRT-PCR (peak levels of viral genomic equivalents). | From baseline (Day -2 or -1) and daily from Day 2 through Day 8
Duration of virus shed into NP swabs post-challenge using qRT-PCR (total numbers of days PCR positive post-challenge). | From baseline (Day -2 or -1) and daily from Day 2 through Day 8

OTHER OUTCOMES:
Baseline and post-challenge neuraminidase inhibition (NAI) antibody GMTs from serum | Baseline (Day -2), and on Days 8, 29, and 61.
Percentage achieving NAI seroconversion (defined as either a pre-challenge titer of <1:10 and post challenge titer greater than or equal to 1:40 or a pre-challenge titer greater than or equal to 1:10 and a four fold rise in post-challenge antibody titer | Baseline (Day -2), and on Days 8, 29, and 61.
Spearman correlations between baseline A/Bethesda/MM2/H2N1 NAI antibody GMT and post challenge total AUC of NP viral shedding measured by qRT-PCR | Baseline (Day -2) and on Days 2-8, 15, 29, and 61
Spearman correlations between baseline A/Bethesda/MM2/H1N1 NAI antibody GMT and post-challenge FLU PRO illness scores | Baseline (Day -2) and Days 2 through Day 14.
Positive, GMT responses for A/Texas/71/2017 (H3N2)-specific sIgA, nonnormalized and normalized for total IgA content in NP swabs | Baseline (Day -2) and Days 8, 29, and 61
Determine the frequency of HLA class I and II alleles as measured by genetic testing | Day 61
To assess the correlation of subject HLA class I and II alleles with development of Mild-to-Moderate Influenza Disease (MMID) post-challenge, pre-existing immune status, and magnitude and breadth of the elicited immune responses post challenge | Days 2 through 8 post-challenge
Summarize the data on systemic and mucosal cytokines induced by challenge and study their relationships to the number of days of persistent influenza infection by PCR. | Baseline (Day -2) pre-challenge through Day 8 post-challenge
Magnitude of influenza-specific T cell responses in circulating Peripheral Blood Mononuclear Cells (PBMC) to conserved T cell epitopes and inactivated virus | Baseline (Day -2) pre-challenge and on Days 4, 6, 8, 15, 29, and 61
Positive, Geometric Mean Fold Rise (GMFR) responses for A/Texas/71/2017 (H3N2)-specific sIgA, nonnormalized and normalized for total IgA content in NP swabs. | Baseline (Day -2) and Days 8, 29, and 61.
Summarize the data on systemic and mucosal cytokines induced by challenge and study their relationships to the number of days of other disease outcomes by PCF. | Baseline (Day -2) pre-challenge through Day 8 post-challenge
Summarize the data on systemic and mucosal cytokines induces by challenge and study their relationships to the number of days of HAI-MN-NAI seroconversion. | Baseline (Day -2) pre-challenge through Day 8 post-challenge

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hoft, MD, PhD, Principal Investigator — Saint Louis University Center for Vaccine Development
Locations (1):
- Saint Louis University Center for Vaccine Development, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study that will generate data for larger studies in the future for which IPD would be shared.

REFERENCES:
- [Background] 22. Centers for Disease Control and Prevention. People at High Risk For Flu Complications. Available at: https://www.cdc.gov/flu/highrisk/index.htm. Accessed 14 February 2025.
- [Background] Friedman J, Hastie T, Tibshirani R. Regularization Paths for Generalized Linear Models via Coordinate Descent. J Stat Softw. 2010;33(1):1-22. PMID 20808728
- [Background] Hasing ME, Hazes B, Lee BE, Preiksaitis JK, Pang XL. A next generation sequencing-based method to study the intra-host genetic diversity of norovirus in patients with acute and chronic infection. BMC Genomics. 2016 Jul 1;17:480. doi: 10.1186/s12864-016-2831-y. PMID 27363999
- [Background] Powers JH, Guerrero ML, Leidy NK, Fairchok MP, Rosenberg A, Hernandez A, Stringer S, Schofield C, Rodriguez-Zulueta P, Kim K, Danaher PJ, Ortega-Gallegos H, Bacci ED, Stepp N, Galindo-Fraga A, St Clair K, Rajnik M, McDonough EA, Ridore M, Arnold JC, Millar EV, Ruiz-Palacios GM. Development of the Flu-PRO: a patient-reported outcome (PRO) instrument to evaluate symptoms of influenza. BMC Infect Dis. 2016 Jan 5;16:1. doi: 10.1186/s12879-015-1330-0. PMID 26729246
- [Background] 18. Food and Drug Administration. Highlights of Prescribing Information. Available at: https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/210854s000lbl.pdf. Accessed 14 February 2025.
- [Background] Kaji M, Watanabe A, Aizawa H. Differences in clinical features between influenza A H1N1, A H3N2, and B in adult patients. Respirology. 2003 Jun;8(2):231-3. doi: 10.1046/j.1440-1843.2003.00457.x. PMID 12753540
- [Background] Shetty N, Shephard MJ, Rockey NC, Macenczak H, Traenkner J, Danzy S, Vargas-Maldonado N, Arts PJ, Le Sage V, Anderson EJ, Lyon GM, Fitts EC, Gulick DA, Mehta AK, El-Chami MF, Kraft CS, Wigginton KR, Lowen AC, Marr LC, Rouphael NG, Lakdawala SS. Influenza virus infection and aerosol shedding kinetics in a controlled human infection model. J Virol. 2024 Dec 17;98(12):e0161224. doi: 10.1128/jvi.01612-24. Epub 2024 Nov 26. PMID 39589151
- [Background] Ortiz JR, Bernstein DI, Hoft DF, Woods CW, McClain MT, Frey SE, Brady RC, Bryant C, Wegel A, Frenck RW, Walter EB, Abate G, Williams SR, Atmar RL, Keitel WA, Rouphael N, Memoli MJ, Makhene MK, Roberts PC, Neuzil KM. A Multicenter, Controlled Human Infection Study of Influenza A(H1N1)pdm09 in Healthy Adults. J Infect Dis. 2023 Aug 11;228(3):287-298. doi: 10.1093/infdis/jiad021. PMID 36702771
- [Background] Memoli MJ, Shaw PA, Han A, Czajkowski L, Reed S, Athota R, Bristol T, Fargis S, Risos K, Powers JH, Davey RT Jr, Taubenberger JK. Evaluation of Antihemagglutinin and Antineuraminidase Antibodies as Correlates of Protection in an Influenza A/H1N1 Virus Healthy Human Challenge Model. mBio. 2016 Apr 19;7(2):e00417-16. doi: 10.1128/mBio.00417-16. PMID 27094330
- [Background] Memoli MJ, Czajkowski L, Reed S, Athota R, Bristol T, Proudfoot K, Fargis S, Stein M, Dunfee RL, Shaw PA, Davey RT, Taubenberger JK. Validation of the wild-type influenza A human challenge model H1N1pdMIST: an A(H1N1)pdm09 dose-finding investigational new drug study. Clin Infect Dis. 2015 Mar 1;60(5):693-702. doi: 10.1093/cid/ciu924. Epub 2014 Nov 20. PMID 25416753
- [Background] Ison MG, Campbell V, Rembold C, Dent J, Hayden FG. Cardiac findings during uncomplicated acute influenza in ambulatory adults. Clin Infect Dis. 2005 Feb 1;40(3):415-22. doi: 10.1086/427282. Epub 2005 Jan 10. PMID 15668866
- [Background] Barroso L, Treanor J, Gubareva L, Hayden FG. Efficacy and tolerability of the oral neuraminidase inhibitor peramivir in experimental human influenza: randomized, controlled trials for prophylaxis and treatment. Antivir Ther. 2005;10(8):901-10. PMID 16430195
- [Background] Waldock J, Cox RJ, Chiu C, Subbarao K, Wildfire A, Barclay W, van Kasteren PB, McCauley J, Russell CA, Smith D, Thwaites RS, Tregoning JS, Engelhardt OG. Inno4Vac Workshop Report Part 1: Controlled Human Influenza Virus Infection Model (CHIVIM) Strain Selection and Immune Assays for CHIVIM Studies, November 2021, MHRA, UK. Influenza Other Respir Viruses. 2024 Nov;18(11):e70014. doi: 10.1111/irv.70014. PMID 39496425
- [Background] Carrat F, Vergu E, Ferguson NM, Lemaitre M, Cauchemez S, Leach S, Valleron AJ. Time lines of infection and disease in human influenza: a review of volunteer challenge studies. Am J Epidemiol. 2008 Apr 1;167(7):775-85. doi: 10.1093/aje/kwm375. Epub 2008 Jan 29. PMID 18230677
- [Background] Taaffe J, Ostrowsky JT, Mott J, Goldin S, Friede M, Gsell P, Chadwick C. Advancing influenza vaccines: A review of next-generation candidates and their potential for global health impact. Vaccine. 2024 Dec 2;42(26):126408. doi: 10.1016/j.vaccine.2024.126408. Epub 2024 Oct 5. PMID 39369576
- [Background] 7. Guidance for Industry. Clinical Data Needed to Support the Licensure of Seasonal Inactivated Influenza Vaccines. U.S. DHHS, FDA, CBER, May 2007.
- [Background] Erbelding EJ, Post DJ, Stemmy EJ, Roberts PC, Augustine AD, Ferguson S, Paules CI, Graham BS, Fauci AS. A Universal Influenza Vaccine: The Strategic Plan for the National Institute of Allergy and Infectious Diseases. J Infect Dis. 2018 Jul 2;218(3):347-354. doi: 10.1093/infdis/jiy103. PMID 29506129
- [Background] 5. COVID-19. Available at https://cepi.net/COVID-19. Accessed 13 February 2025.
- [Background] 2. CDC Seasonal Flu Vaccine Effectiveness Studies. Available at https://www.cdc/gpv/flu-vaccines-work/php/effectiveness-studies/index,html. Accessed 13 February 2025.
- [Background] Mao T, Israelow B, Pena-Hernandez MA, Suberi A, Zhou L, Luyten S, Reschke M, Dong H, Homer RJ, Saltzman WM, Iwasaki A. Unadjuvanted intranasal spike vaccine elicits protective mucosal immunity against sarbecoviruses. Science. 2022 Nov 25;378(6622):eabo2523. doi: 10.1126/science.abo2523. Epub 2022 Nov 25. PMID 36302057
- [Background] Gagne M, Flynn BJ, Andrew SF, Marquez J, Flebbe DR, Mychalowych A, Lamb E, Davis-Gardner ME, Burnett MR, Serebryannyy LA, Lin BC, Ziff ZE, Maule E, Carroll R, Naisan M, Jethmalani Y, Pessaint L, Todd JM, Doria-Rose NA, Case JB, Dmitriev IP, Kashentseva EA, Ying B, Dodson A, Kouneski K, O'Dell S, Wali B, Ellis M, Godbole S, Laboune F, Henry AR, Teng IT, Wang D, Wang L, Zhou Q, Zouantchangadou S, Van Ry A, Lewis MG, Andersen H, Kwong PD, Curiel DT, Roederer M, Nason MC, Foulds KE, Suthar MS, Diamond MS, Douek DC, Seder RA. Mucosal adenovirus vaccine boosting elicits IgA and durably prevents XBB.1.16 infection in nonhuman primates. Nat Immunol. 2024 Oct;25(10):1913-1927. doi: 10.1038/s41590-024-01951-5. Epub 2024 Sep 3. PMID 39227514
- [Background] Taubenberger JK, Morens DM. The 1918 Influenza Pandemic and Its Legacy. Cold Spring Harb Perspect Med. 2020 Oct 1;10(10):a038695. doi: 10.1101/cshperspect.a038695. PMID 31871232